CLINICAL TRIAL: NCT02188992
Title: Early Prediction of Severe Sepsis (ExPRESSepsis) Study
Brief Title: Early PREdiction of Severe Sepsis I (ExPRES-Sepsis I) Study
Acronym: ExPRES
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Technology Strategy Board, United Kingdom (Other); Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013/0267
Record Dates: First submitted 2014-07-07; First posted 2014-07-14 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2014-07

CONDITIONS: Sepsis
Keywords: Sepsis; Immune activation; Systemic Inflammation; Emergency Medicine; Critical Care
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of serum and plasma will be stored frozen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: Patients with sepsis syndrome, without criteria for severe sepsis/septic shock. These patients are recruited from the emergency department.
- Cohort 2: Patients with community acquired sepsis syndrome REQUIRING critical care admission due to severity of sepsis. These patients are recruited from the critical care areas (ICU/HDU).
- Cohort 3: Patients without sepsis syndrome. Age and gender matched to cohort 1, and recruited from Emergency Department.

SUMMARY:
Between 6 and 16% of patients presenting to hospital emergency departments have infections, with half of these having signs of systemic inflammation (known as 'sepsis'). A second issue is that, at time of presentation, it can be difficult to determine who has inflammation as a result of infection and who does not.

Some of the patients with infections will deteriorate to organ failure ('severe sepsis') including failure of the heart and blood vessels to maintain normal blood pressure ('septic shock'). Septic shock as arguably the most dangerous form of severe sepsis is associated with a significant mortality, which can be reduced by early intervention. However identifying those patients who are at high risk of deteriorating to septic shock can be difficult on initial presentation to hospital, and thus these patients risk being 'triaged' to an inappropriate level of care and/or missing the crucial early interventions which can modify mortality. Equally failure to identify which patients have underlying infections can lead to potential inappropriate targeting of antibiotics. Existing clinical and laboratory tests are often unable to accurately identify those patients with infection, and those who are likely to deteriorate to severe sepsis and septic shock.

Investigators in this group have recently identified several signatures of immune system activation which predict those patients who are likely to deteriorate, and which patients with suspected infection subsequently have this confirmed. Such tests would have major benefits for the management of patients with early suspected infection and sepsis if they can be translated into a test usable in everyday clinical practice. This study aims to determine the prevalence of these markers in a cohort of patients admitted with suspected sepsis, and their predictive ability for developing established septic shock. From this investigators aim to derive an optimal test, to be tested in a validation cohort (ExPRES-Sepsis II) which will be suitable for everyday clinical practice, and thus take the next step towards developing a market-ready test.

Study hypothesis is:

Measurement of markers of immune activation will allow i) Risk stratification for deterioration into severe sepsis ii) Risk stratification for death amongst patients presenting with sepsis iii) Identification of patients with confirmed sepsis

ELIGIBILITY:
Inclusion Criteria:

* Age >16 (>18 in England)
* SIRS criteria met (2 or more of White Cell Count (WCC) >11 or <4, Heart Rate (HR) >90, Respiratory Rate (RR) >20 or temp >38 or <36oC)
* Clinical suspicion of sepsis (cultures taken or antibiotics started)
* Enrolled within 12 hours of hospital admission

Exclusion Criteria:

* Acute pancreatitis
* Septic shock at time of enrolment
* Severe organ failure at time of enrolment (immediate requirement for ventilation, vasopressor or renal replacement therapy)
* Haematological malignancy
* Recent chemotherapy (past 2 weeks)
* Myelodysplastic syndromes
* Known neutropaenia
* HIV infection
* Pregnancy
* Blood transfusion >4 units in past week
* Oral Corticosteroids for >24 hours prior to enrolment
* Decision not for active therapy/ palliative care at admission
* Lacking in capacity to consent and nearest relative/welfare guardian not available for consultation and proxy consent (Scotland only)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the initial 12 hours following presentation to hospital with suspected sepsis, i.e. patients with signs of systemic inflammation (i.e. meeting criteria for SIRS) where the treating clinician takes microbial samples and/or starts empiric antibiotics.
Sampling Method: Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Development of septic shock | Within first 72 hours
Confirmation of suspected infection | within first 72 hours

SECONDARY OUTCOMES:
Hospital outcome (lived/died) | Within first 72 hours
Time to septic shock onset | Within the first 72 hours
Death from sepsis | Within first 72 hours
Organ dysfunction, total and individual organs as determined by SOFA score | within first 72 hours
subsequent admission to critical care | within first 72 hours
Changes in immune activation in those patients who develop any of the events mention in previous outcomes (i.e. septic shock, death, organ dysfunction, admission to critical care) | within first 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tim S Walsh, MD, Principal Investigator — NHS Lothian/University of Edinburgh; John Wright, MD, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust; Manu Shankar-Hari, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Andrew Conway Morris, MD, Principal Investigator — University of Cambridge; John Simpson, MD, Principal Investigator — Newcastle University; Alasdair Gray, MD, Principal Investigator — NHS Lothian/University of Edinburgh
Locations (3):
- United Kingdom (3):
  - Royal Infirmary of Edinburgh, Edinburgh
  - St Thomas' Hospital, London
  - Royal Victoria Infirmary, Newcastle

REFERENCES:
- [Derived] Shankar-Hari M, Datta D, Wilson J, Assi V, Stephen J, Weir CJ, Rennie J, Antonelli J, Bateman A, Felton JM, Warner N, Judge K, Keenan J, Wang A, Burpee T, Brown AK, Lewis SM, Mare T, Roy AI, Wright J, Hulme G, Dimmick I, Gray A, Rossi AG, Simpson AJ, Conway Morris A, Walsh TS. Early PREdiction of sepsis using leukocyte surface biomarkers: the ExPRES-sepsis cohort study. Intensive Care Med. 2018 Nov;44(11):1836-1848. doi: 10.1007/s00134-018-5389-0. Epub 2018 Oct 5. PMID 30291379
- [Derived] Datta D, Conway Morris A, Antonelli J, Warner N, Brown KA, Wright J, Simpson AJ, Rennie J, Hulme G, Lewis SM, Mare TA, Cookson S, Weir CJ, Dimmick I, Keenan J, Rossi AG, Shankar-Hari M, Walsh TS; ExPRES Sepsis Investigators. Early PREdiction of Severe Sepsis (ExPRES-Sepsis) study: protocol for an observational derivation study to discover potential leucocyte cell surface biomarkers. BMJ Open. 2016 Aug 1;6(8):e011335. doi: 10.1136/bmjopen-2016-011335. PMID 27481622